CLINICAL TRIAL: NCT01143181
Title: A Multicenter, Open-label Study of CMX001 Treatment of Serious Diseases or Conditions Caused by Double-stranded DNA Viruses
Brief Title: Study to Assess Brincidofovir Treatment of Serious Diseases or Conditions Caused by Double-stranded DNA Viruses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMX001-350
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Double-stranded DNA Virus
Keywords: Cytomegalovirus; Adenovirus; Herpes simplex virus; Vaccinia virus; Variola virus
MeSH Terms: conditions — Adenoviridae Infections; Herpes Simplex; Vaccinia; Smallpox | interventions — brincidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brincidofovir (Experimental): Subjects received either a weight-based or a fixed-dose of oral brincidofovir (BCV) once weekly or twice weekly for up to 3 months until clinical disease was resolved or stabilized and/or viral DNA polymerase chain reaction testing was negative for 4 consecutive weeks, whichever was longer.
  Interventions: Drug: Brincidofovir

INTERVENTIONS:
Drug: Brincidofovir — Brincidofovir (BCV) was administered orally either once or twice weekly for up to 3 months. Treatment may have been extended for an additional 3 months depending a satisfactory review of safety parameters. Subjects could not receive more than a total of 6 months of treatment with BCV without prior approval.
  Other Names: CMX001; BCV

SUMMARY:
This was a multicenter, open-label study of oral brincidofovir (BCV) treatment of serious disease or conditions caused by double-stranded DNA (dsDNA) virus(es). Subjects received either a weight-based or a fixed dose of oral BCV once weekly (QW) or twice weekly (BIW) for up to 3 months until clinical disease was resolved or stabilized and/or viral DNA by polymerase chain reaction testing was negative for 4 consecutive weeks, whichever was longer. Under the first protocol amendment, adults and adolescents (≥13 years) received 200 mg or 300 mg BCV BIW (not to exceed 4 mg/kg total weekly dose) depending on the difficulty of treating their disease (i.e., Group 1 or Group 2, respectively), and pediatric subjects (≤12 years) received 4 mg/kg BCV BIW. Under the second protocol amendment, adults and adolescents (≥13 years), regardless of viral infection/disease, had a maximum weekly dose of 200 mg, i.e., 200 mg QW or 100 mg BIW; not to exceed 4mg/kg total weekly dose. Pediatric subjects (≤12 years), regardless of viral infection/disease, had a maximum weekly dose of 4 mg/kg, i.e., 4 mg/kg QW or 2 mg/kg BIW; not to exceed 200 mg.

DETAILED DESCRIPTION:
This was a multicenter, open-label study of oral brincidofovir (BCV) treatment of serious disease or conditions caused by double-stranded DNA (dsDNA) virus(es).

Subjects with a life-threatening or serious disease or condition caused by infection with any dsDNA virus(es), who met the protocol eligibility criteria and who were approved by the Chimerix Medical Monitor were enrolled in this open-label treatment study. During the course of the study, the viral disease indications were narrowed in Amendment 2 to cytomegalovirus, adenovirus, herpes simplex virus, vaccinia virus, variola virus, or monkeypox virus to focus on indications that were under study in controlled clinical trials of oral BCV and on viral disease with few, if any, options for treatment. However, subjects with other viral disease indications may have been enrolled with the approval of the Chimerix Medical Monitor.

Subjects received either a weight-based or a fixed dose of oral BCV once weekly (QW) or twice weekly (BIW) for up to 3 months until clinical disease was resolved or stabilized and/or viral DNA by polymerase chain reaction testing was negative for 4 consecutive weeks, whichever was longer. Subjects who met criteria for resolution of viral disease may have: 1) discontinued BCV; 2) reduced the dose or dosing frequency of BCV; or 3) continued BCV QW or BIW, depending on the investigator's assessment of the risk of relapse and following discussion with the Chimerix medical monitor.

ELIGIBILITY:
Inclusion Criteria

Subjects were required to meet all of the following inclusion criteria in order to participate in the study:

1. Had an immediately life-threatening or serious disease or condition caused by infection with a double-stranded DNA virus (including subjects with recurrent viral disease). [Note: During the course of the study, the viral disease indications were narrow to focus on indications that were under study in controlled clinical trials of brincidofovir (BCV) and on viral diseases that had few, if any, options for treatment, including cytomegalovirus (CMV), adenovirus (AdV), herpes simplex virus (HSV), vaccinia virus (VAVC), variola virus (VARV) or monkeypox viruses(s).]
2. Had a life expectancy of at least 2 weeks and commitment to continuation of supportive care for at least 4 weeks.
3. Were able to ingest and absorb oral medication (in the judgment of the investigator and based on lack of significant gastrointestinal [GI] pathology such as small bowel resection or ileus). [Note: Use of total parenteral nutrition was not in and of itself exclusionary as long as the reason for use did not disqualify the subject based on this criterion.]
4. Were willing and able to understand and provide written informed consent. [Note: For minors or those incapable of providing written informed consent (i.e., incapacitated), consent was provided by a parent or legal guardian or representative who could understand and provide written informed consent.]
5. Were willing and able, to the best of his or her (or parent/guardian) knowledge, to participate in all required study activities for the duration of the study.
6. If female of reproductive potential, agreed to use 2 acceptable methods of birth control throughout the study with at least 1 being a barrier method.
7. In the judgment of the investigator, subjects for whom no comparable or satisfactory therapeutic alternative was available

Exclusion Criteria

Subjects were not to be enrolled if they met any of the following exclusion criteria:

1. Were pregnant or currently nursing.
2. Had hypersensitivity to cidofovir or BCV.
3. Had a long-term prognosis that included a poor likelihood of survival due to irreversible organ failure including, for example, subjects with frank hepatic failure and adults with Grade 4 graft versus host disease of the GI tract.
4. Were eligible for enrollment and able to participate in a clinical trial evaluating BCV. [Note: Per the FDA guidance, subjects eligible and able to participate in a controlled clinical study evaluating BCV were not eligible for participation in this study. Subjects who did not meet eligibility criteria for a controlled BCV clinical study or who were unable to participate because, for example, of logistical or other issues were eligible to participate in this study. The investigator verified that his/her subjects met this criterion on the Eligibility electronic case report form. A subject simply preferring enrollment in this study over a BCV controlled clinical trial did not qualify for enrollment in this study.]
5. Had any other condition that would have, in the judgment of the investigator, put the subject at increased risk during participation in the study or interfered with the conduct of the study.
6. Had a serum total bilirubin value >5 x the upper limit of normal reference range, taking into account the age and/or gender of the subject. [Note: In order to avoid any unwarranted delay to the start of BCV treatment, compliance with this exclusion criterion may have been determined based on the results of testing performed at a local safety laboratory, rather than waiting for results from the designated central safety laboratory. If relying on local safety laboratory test results, the blood sample must have been collected no more than 7 days prior to the scheduled first dose administration on Day 0, otherwise it was repeated. A subject whose elevated bilirubin was due to the underlying viral disease may still have been enrolled into the study if the participation of the subject was prospectively approved by the Chimerix Medical Monitor.]

Subjects with acute or chronic renal impairment, pediatric and adolescent subjects, and subjects aged 65 years and older were included in this study. Subjects with hepatic impairment were included unless the investigator judged that the subject had irreversible hepatic compromise.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (37):
  - Loma Linda University Hospital, Loma Linda, California
  - Children's Hospital of LA, Los Angeles, California
  - UCLA Department of Medicine, Los Angeles, California
  - CHOC Children's, Orange, California
  - Univeristy of San Francisco, San Francisco, California
  - Lucile Packard Children's Hospital, Stanford, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Childrens Hospital LSU, New Orleans, Louisiana
  - NIH, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mt. Sinai, New York, New York
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Institute, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Levine Children's Hospital Carolina Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
  - Intermountain BMT program LDS Hospital, Salt Lake City, Utah
  - University of Washington-Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Tippin TK, Morrison ME, Brundage TM, Mommeja-Marin H. Brincidofovir Is Not a Substrate for the Human Organic Anion Transporter 1: A Mechanistic Explanation for the Lack of Nephrotoxicity Observed in Clinical Studies. Ther Drug Monit. 2016 Dec;38(6):777-786. doi: 10.1097/FTD.0000000000000353. PMID 27851688

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an expanded access study with the primary objective of providing brincidofovir (BCV) to subjects with serious or life-threatening conditions caused by double-stranded DNA viral infections. All subjects enrolled received BCV for up to 3 months until their clinical disease was resolved or stabilized and/or viral DNA testing was negative for 4 consecutive weeks, whichever was longer.
Groups:
- BCV (≤4 mg/kg/Week); BCV (>4 mg/kg/Week): Pediatric subjects (≤12 years) who received BCV once or twice weekly.
- BCV (≤200 mg/Week); BCV (>200 mg/Week): Adult/adolescent subjects (≥13 years) who received BCV once or twice weekly.
Period: Overall Study
Arm/Group | BCV (≤4 mg/kg/Week) | BCV (>4 mg/kg/Week) | BCV (≤200 mg/Week) | BCV (>200 mg/Week)
Started | 30 | 38 | 102 | 40
Completed | 14 | 22 | 58 | 17
Not Completed | 16 | 16 | 44 | 23

BASELINE CHARACTERISTICS:
Population: This was an expanded access study with the primary objective of providing brincidofovir (BCV) to subjects with serious or life-threatening conditions caused by double-stranded DNA viral infections. All subjects enrolled received BCV for up to 3 months until their clinical disease was resolved or stabilized and/or viral DNA testing was negative for 4 consecutive weeks, whichever was longer.
Groups:
- Total: Total of all reporting groups
Arm/Group | BCV (≤4 mg/kg/Week) | BCV (>4 mg/kg/Week) | BCV (≤200 mg/Week) | BCV (>200 mg/Week) | Total
Number analyzed (Participants) | 30 | 38 | 102 | 40 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.2 (2.68) | 5.9 (3.70) | 45.3 (17.21) | 45.7 (17.57) | 32.5 (23.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 41 | 18 | 87
  Male | 16 | 24 | 61 | 22 | 123

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Had a Sustained and Significant Reduction in Plasma Viral Load of Primary dsDNA Virus
Description: Proportion of subjects who achieved a confirmed reduction in viral load for the primary dsDNA virus of ≥1 log10 copies/mL from baseline or to an undetectable level. Confirmation required the reduction in viral load (i.e., decrease of ≥ 1 log10 copies/mL from baseline or to undetectable levels) to be maintained at the next assessment for the subject to be considered a success.
Time Frame: 3 months
Population: Only subjects who achieved a confirmed reduction in viral load for the primary dsDNA virus of ≥1 log10 copies/mL from baseline or to an undetectable level were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | BCV (≤4 mg/kg/Week) | BCV (>4 mg/kg/Week) | BCV (≤200 mg/Week) | BCV (>200 mg/Week)
Number analyzed (Participants) | 25 | 28 | 79 | 28
Participants | 15 | 18 | 39 | 13

ADVERSE EVENTS:
Arm/Group | BCV (≤4 mg/kg/Week) | BCV (>4 mg/kg/Week) | BCV (≤200 mg/Week) | BCV (>200 mg/Week)
Serious Adverse Events (participants affected / at risk) | 27/30 | 32/38 | 80/102 | 35/40
Other Adverse Events (participants affected / at risk) | 30/30 | 37/38 | 101/102 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BCV (≤4 mg/kg/Week) (N=30) | BCV (>4 mg/kg/Week) (N=38) | BCV (≤200 mg/Week) (N=102) | BCV (>200 mg/Week) (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 4 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 9 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 3 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 4 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dental discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 17 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1 | 2
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Malabsorption (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 9 | 4
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 7 | 4
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 1 | 0
Multi-organ failure (General disorders) | 3 | 1 | 7 | 6
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 5 | 6 | 11 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholestatic liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 3 | 0
Venooclusive liver disease (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Acute graft versus host disease (Immune system disorders) | 0 | 2 | 13 | 7
Chronic graft versus host disease (Immune system disorders) | 3 | 1 | 4 | 2
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 1
Immune reconstitution syndrome (Immune system disorders) | 0 | 0 | 1 | 0
Lung transplant rejection (Immune system disorders) | 0 | 0 | 0 | 1
Adenoviral hepatitis (Infections and infestations) | 1 | 0 | 1 | 0
Adenovirus infection (Infections and infestations) | 1 | 1 | 0 | 0
Aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0
BK virus infection (Infections and infestations) | 0 | 1 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 3 | 1
Bronchiectasis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0
Central nervous system infection (Infections and infestations) | 0 | 0 | 1 | 0
Citrobacter infection (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 2 | 3
Corona virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 0 | 1
Disseminated cytomegaloviral infection (Infections and infestations) | 0 | 0 | 1 | 0
Encephalitis herpes (Infections and infestations) | 0 | 0 | 1 | 0
Enterobacter infection (Infections and infestations) | 0 | 0 | 1 | 0
Enterobacter pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Enterobacter sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 2 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Fungal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Human herpesvirus 6 infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
JC virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 2 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 2 | 0
Legionella infection (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 1 | 2 | 0
Meningoencephalitis adenoviral (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 2 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia adenoviral (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 3 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia herpes viral (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 0 | 2 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0 | 3 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 2 | 1
Septic shock (Infections and infestations) | 0 | 1 | 2 | 1
Serratia infection (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis fungal (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 2 | 1 | 3 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 2 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 0 | 1 | 0
Stenotrophomonas sepsis (Infections and infestations) | 1 | 1 | 2 | 0
Toxoplasmosis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Zygomycosis (Infections and infestations) | 0 | 0 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood stem cell transplant failure (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Transplant failure (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 3 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 3 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
Pancreatic enzymes increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 6 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Adult T-cell lymphoma/leukaemia refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 1
Embolic cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 2 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 3 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 2 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2 | 4 | 4
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 2 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5 | 1
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 9 | 4
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 4 | 7 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 2 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0
Venous stenosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCV (≤4 mg/kg/Week) (N=30) | BCV (>4 mg/kg/Week) (N=38) | BCV (≤200 mg/Week) (N=102) | BCV (>200 mg/Week) (N=40)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 5 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 16 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 10 | 3
Bradycardia (Cardiac disorders) | 2 | 3 | 2 | 1
Pericardial effusion (Cardiac disorders) | 2 | 2 | 2 | 1
Tachycardia (Cardiac disorders) | 2 | 1 | 9 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 2 | 2 | 2
Dry eye (Eye disorders) | 1 | 0 | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 7 | 26 | 4
Ascites (Gastrointestinal disorders) | 1 | 3 | 5 | 3
Colitis (Gastrointestinal disorders) | 0 | 3 | 5 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 8 | 2
Diarrhoea (Gastrointestinal disorders) | 12 | 22 | 61 | 19
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 3 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 6 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 4 | 1 | 3
Haematochezia (Gastrointestinal disorders) | 1 | 2 | 2 | 1
Ileus (Gastrointestinal disorders) | 2 | 1 | 1 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 6 | 42 | 9
Pancreatitis (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Pneumatosis (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Vomiting (Gastrointestinal disorders) | 8 | 13 | 30 | 7
Asthenia (General disorders) | 0 | 0 | 3 | 3
Chest pain (General disorders) | 0 | 0 | 0 | 3
Chills (General disorders) | 1 | 1 | 7 | 2
Fatigue (General disorders) | 1 | 1 | 13 | 1
Generalized oedema (General disorders) | 2 | 1 | 6 | 0
Muscosal inflammation (General disorders) | 2 | 1 | 0 | 0
Multi-organ failure (General disorders) | 3 | 1 | 7 | 6
Oedema peripheral (General disorders) | 0 | 1 | 17 | 2
Pain (General disorders) | 1 | 2 | 3 | 0
Pyrexia (General disorders) | 13 | 9 | 25 | 4
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 2
Hepatic failure (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 7 | 3
Acute graft versus host disease (Immune system disorders) | 8 | 11 | 30 | 11
Chronic graft versus host disease (Immune system disorders) | 3 | 2 | 8 | 3
Adenovirus infection (Infections and infestations) | 2 | 1 | 2 | 0
BK virus infection (Infections and infestations) | 1 | 2 | 4 | 2
Bacteraemia (Infections and infestations) | 2 | 2 | 2 | 1
Candidiasis (Infections and infestations) | 0 | 4 | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 3 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 3 | 6 | 5
Cytomegalovirus colitis (Infections and infestations) | 2 | 0 | 1 | 1
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0 | 3 | 2
Enterococcal sepsis (Infections and infestations) | 0 | 1 | 1 | 2
Epstein-Barr viraemia (Infections and infestations) | 0 | 0 | 6 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 2 | 0 | 0
Human herpesvirus 6 infection (Infections and infestations) | 2 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 2 | 2
Oral candidiasis (Infections and infestations) | 1 | 2 | 6 | 0
Pneumonia (Infections and infestations) | 3 | 3 | 4 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 3 | 0 | 2 | 2
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0 | 4 | 2
Sinusitis (Infections and infestations) | 1 | 2 | 2 | 2
Staphylococcal bacteraemia (Infections and infestations) | 2 | 1 | 6 | 2
Systemic candida (Infections and infestations) | 0 | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 3 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 0
Transplant failure (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 4 | 17 | 6
Aspartate aminotransferase increased (Investigations) | 5 | 3 | 17 | 4
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 8 | 0
Blood bilirubin increased (Investigations) | 2 | 4 | 4 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 8 | 1
Clostridium test positive (Investigations) | 1 | 0 | 2 | 2
Neutrophil count decreased (Investigations) | 4 | 2 | 4 | 0
Weight decreased (Investigations) | 1 | 1 | 6 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 7 | 17 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 8 | 3
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 3 | 3
Fluid retention (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 9 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 4 | 9 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 1 | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 8 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 8 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 8 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 6 | 0
Epstein-Barr virus associated lymphoproliferative (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3 | 3
Convulsion (Nervous system disorders) | 1 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 6 | 3
Encephalopathy (Nervous system disorders) | 0 | 1 | 3 | 3
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 3 | 12 | 3
Tremor (Nervous system disorders) | 0 | 1 | 7 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 6 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 6 | 4
Anxiety (Psychiatric disorders) | 2 | 2 | 6 | 3
Confusional state (Psychiatric disorders) | 0 | 0 | 8 | 1
Depression (Psychiatric disorders) | 2 | 0 | 6 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 5 | 3
Mental status changes (Psychiatric disorders) | 2 | 0 | 8 | 2
Haematuria (Renal and urinary disorders) | 0 | 2 | 4 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 6 | 6 | 4
Renal failure (Renal and urinary disorders) | 4 | 3 | 4 | 4
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 16 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 14 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 7 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 8 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 8 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 10 | 2
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 3 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 10 | 6
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 6 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 3 | 10 | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2
Hypertension (Vascular disorders) | 8 | 3 | 7 | 4
Hypotension (Vascular disorders) | 6 | 7 | 16 | 5
Hypovolaemic shock (Vascular disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 18 months after the end of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given opportunity to review and comment. Institution publications may be delayed up to an additional 60 days to allow Sponsor to seek patent protection.